CLINICAL TRIAL: NCT06831786
Title: Immunogenicity to SARS-CoV-2 of Co-administering Bivalent mRNA BNT162b2 Booster and Quadrivalent Influenza Vaccine Among Healthy Volunteers: A Pilot Study
Brief Title: Immunogenicity of COVID-19 Vaccine Co-administration With Influenza Vaccine in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sarunyou Chusri, Principal Investigator, Clinical Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REC.66-462-14-1
Record Dates: First submitted 2025-02-15; First posted 2025-02-18 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: COVID - 19
Keywords: co-administration; immunogenicity; cell-medicated immune response; influenza vaccine; COVID-19 vaccine; SARS-CoV-2 vaccine
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bivalent mRNA BNT162b2 (Active Comparator): Administering a booster dose of the bivalent mRNA vaccine BNT162b2.
  Interventions: Biological: Bivalent mRNA SARS-CoV-2 vaccine
- Quardrivalent influenza vaccine (Experimental): Administering a VaxigripTetra™
  Interventions: Biological: Quardrivalent influenza vaccine
- Co-administration (Experimental): Co-administering bivalent mRNA vaccine BNT162b2 and VaxigripTetra™
  Interventions: Biological: Bivalent mRNA SARS-CoV-2 vaccine; Biological: Quardrivalent influenza vaccine

INTERVENTIONS:
Biological: Bivalent mRNA SARS-CoV-2 vaccine — Administering a booster dose of the bivalent mRNA vaccine BNT162b2
  Arms: Bivalent mRNA BNT162b2; Co-administration
Biological: Quardrivalent influenza vaccine — Administering a VaxigripTetra™
  Arms: Co-administration; Quardrivalent influenza vaccine

SUMMARY:
This study, a pilot randomized controlled trial, single-blind (outcome assessor), evaluating the immune response (both humoral and cell-mediated) against SARS-CoV-2 and the safety of three different vaccine administration approaches: the SARS-CoV-2 mRNA vaccine alone, the influenza vaccine alone, and the co-administration of both vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Thai adults aged 18-60 years, who have vaccinated COVID-19 and influenza vaccine more than 6 months.
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 1-month follow-up of the study.
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator and meet the requirements of immunization.
* The subject can provide with informed consent and sign informed consent form (ICF).

Exclusion Criteria:

* Have history of influenza or COVID-19 infection within 6 months.
* Have the medical history or family history of convulsion, epilepsy, encephalopathy, and psychosis.
* Be allergic to any component of the research vaccines or used to have a history of hypersensitivity or serious reactions to vaccination.
* History of Guillain-Barré syndrome.
* Women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan within six months of after baseline period.
* Have infectious diseases, including HIV and SARS-CoV-2 infection or any symptom of common cold.
* Have history of SARS-CoV-2 infection less than 6 months.
* Having severe chronic diseases or condition in progress cannot be controlled. For example, poor controlled DM and uncontrolled HT.
* Have the history of urticaria 1 year before receiving the investigational vaccine.
* Have known underlying diseases of thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection).
* Having needle sickness.
* Have the history of immunosuppressive therapy, cytotoxic therapy, or systemic corticosteroids.
* Have received blood products within 4 months before injection of investigational vaccines.
* Under anti-tuberculosis treatment.
* Not be able to follow the protocol, or not be able to understand the informed consent according to the researcher's judgment, due to various medical, psychological, social, or other conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarunyou Chusri, M.D., Ph.D., Principal Investigator — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
The data will be kept anonymized.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited between March and April 2024 at Songklanagarind Hospital, Faculty of Medicine, Prince of Songkla University, Hat Yai, Thailand.
Pre-assignment Details: A total of 42 adults were screened for eligibility. Six were excluded because of uncontrolled chronic diseases, leaving 36 participants who were randomized.
Groups:
- COVID-19 vaccine: Administering a booster dose of the bivalent mRNA vaccine BNT162b2 and evaluate immune response against SARS-CoV-2 at baseline and 4 week post-vaccination
- Influenza vaccine: Administering a VaxigripTetra™ and evaluate immune response against SARS-CoV-2 at baseline and 4 week post-vaccination
- Co-administration: Co-administering bivalent mRNA vaccine BNT162b2 and VaxigripTetra™, then evaluate immune response against SARS-CoV-2 at baseline and 4 week post-vaccination
Period: Overall Study
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
Started (Day 0 of vaccination) | 12 | 12 | 12
Completed (4 weeks post vaccination) | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID-19 Vaccine | Influenza Vaccine | Co-administration | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 28 [25 to 38] | 39 [25 to 41] | 29 [25 to 41] | 31 [25 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 8 | 26
  Male | 2 | 4 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration from last COVID-19 vaccination [Median (Inter-Quartile Range); unit: week] — Duration from last COIVD-19 vaccine dose, any type of vaccines
  week | 90 [85 to 110.25] | 85.5 [81.5 to 105] | 85.5 [59 to 96.25] | 87.5 [82 to 107]

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean (GM) of Interferon-gamma (IFN-γ) Response Against the SARS-CoV-2 Virus at Baseline
Description: IFN-γ response against the SARS-CoV-2 virus, measured by the ELISpot assay
Time Frame: Before vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: SFCs/10⁶ PBMCs
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
Number analyzed (Participants) | 12 | 12 | 12
SFCs/10⁶ PBMCs | 19.6 [8.8 to 43.9] | 14 [4.6 to 42.7] | 12.6 [6.5 to 24.7]

2. Primary Outcome: Geometric Mean (GM) of Interferon-gamma (IFN-γ) Response Against the SARS-CoV-2 Virus at 4 Weeks
Description: IFN-γ response against the SARS-CoV-2 virus, measured by the ELISpot assay
Time Frame: 4 weeks post vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: SFCs/10⁶ PBMCs
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
Number analyzed (Participants) | 12 | 12 | 12
SFCs/10⁶ PBMCs | 59.9 [26.2 to 136.9] | 15.2 [4.5 to 51] | 61.6 [37.1 to 102.2]

3. Primary Outcome: Geometric Mean (GM) of IgG Response Against the SARS-CoV-2 Virus at Baseline
Description: IgG response against the SARS-CoV-2 virus, measured by ELISA.
Time Frame: before vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/mL
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
Number analyzed (Participants) | 12 | 12 | 12
BAU/mL | 1276.3 [933.9 to 1744.1] | 1074.2 [574.3 to 2009.3] | 1299.7 [729.7 to 2314.8]

4. Primary Outcome: Geometric Mean (GM) of IgG Response Against the SARS-CoV-2 Virus at 4 Weeks
Description: IgG response against the SARS-CoV-2 virus, measured by ELISA.
Time Frame: 4 weeks post vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/mL
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
Number analyzed (Participants) | 12 | 12 | 12
BAU/mL | 10456.1 [7688.6 to 14219.7] | 1008.0 [568.9 to 1786.2] | 8558.7 [5666.6 to 12926.9]

ADVERSE EVENTS:
Time Frame: From vaccination until 28 days post vaccination
Description: Pre-specified adverse events included solicited local and systemic reactions, assessed at Day 7 and Day 28 post-vaccination. Unsolicited adverse events were monitored daily from Day 1 through Day 28. Serious adverse events were monitored throughout Days 1-28.
Arm/Group | COVID-19 vaccine | Influenza vaccine | Co-administration
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 10/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-19 vaccine (N=12) | Influenza vaccine (N=12) | Co-administration (N=12)
Redness at injection site (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
pain at injection site (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9) | 10 (10)
swelling at injection site (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
mass at injection site (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 9 (9)
Malaise (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 5 (5)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
fever (Immune system disorders) | 1 (1) | 0 (0) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As a single-center pilot study with a limited number of participants, the findings may not be generalizable. The short follow-up duration also restricts conclusions about long-term safety and immune responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT06831786/Prot_SAP_000.pdf